CLINICAL TRIAL: NCT04363242
Title: A Phase 1 Dose Escalation Trial of SYN125 Single Agent in Solid Tumors and in Combination With Fixed Dose SYN004 in Patients With Epithelial Cancers With EGFR Expressions.
Brief Title: A Study to Find the MTD of SYN125 in People With Solid Tumors and the MTD of SYN125 With a Fixed Dose of SYN004 in People in Patients With Epithelial Cancers With EGFR Expressions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synermore Biologics Co., Ltd. (Industry)
Collaborators: Synermore Biologics USA Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYN125-001
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Epithelial Carcinoma; Solid Tumor
Keywords: Epithelial cancer; Epithelial Growth Factor Receptor expression; EGFR
MeSH Terms: conditions — Carcinoma | interventions — SYN-004

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Dose escalation of SYN125. Each dose level (low, medium, high) will be tested in a cohort of 3 patients. If no dose-limiting toxicity (DLT) is observed in the 3 patients, dose escalation will continue to the next SYN125 dose level.
  Interventions: Biological: SYN125
- Part B (Experimental): Dose escalation of SYN125 administered with a fixed-dose of SYN004 (SYN004 will be administered immediately after SYN125 infusion is complete, if tolerated). Once cohorts with low and medium dose levels in Part A are completed and no DLTs are observed per cohort, Part B with the SYN125 low dose level + SYN004 will start and run in parallel with Part A. The high dose of SYN125 in a cohort in Part A will begin along with Part B.
  Interventions: Biological: SYN125; Biological: SYN004

INTERVENTIONS:
Biological: SYN125 — Administered by IV infusion
Biological: SYN004 — Administered by IV infusion
  Arms: Part B

SUMMARY:
A Phase 1 Dose Escalation Trial of SYN125 Single Agent in the Treatment of Solid Tumors and in Combination With Fixed Dose SYN004 in Patients With Cancer of the Internal or External Lining of the Body.

DETAILED DESCRIPTION:
Humans have an immune system that can protect and fight infections and abnormal cells. T-cells are a type of cell produced by the body that can attack and kill cancer cells. Unfortunately, many cancer cells have ways preventing T-cells from working properly. SYN125 and SYN004 can make T-cells work again. This is a study to find the maximum tolerated dose of SYN125 when it is used as a single treatment (Part A) for solid tumors, and when it is used as a combined treatment with a fixed dose of SYN004 (Part B), in patients with epithelial cancers with EGFR (epithelial growth factor receptor) expressions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Have documented diagnosis of recurrent or metastatic solid tumors for whom no standard treatment options are available (Part A only).
* Have epithelial cancers which have endothelial growth factor receptor (EGFR) expressions (not necessarily mutated or over-expressed) (Part B only).

Note: Prior EGFR (epidermal growth factor receptor) therapy and approved checkpoint inhibitor therapy are allowed but not required.

* Prior anti-PD-1 (programmed cell death 1), anti-PD-L1 (programmed death-ligand 1), anti-PD-L2 (programmed death-ligand 2), anti-cytotoxic T-lymphocyte antigen (CTLA-4) are allowed, where the wash-out period will be 28 days from last dose of previous therapy except for palliative RT and smaller molecular oral therapeutic agents where 5 half-lives or 28 days, whichever is shorter, will apply (Part A and Part B).
* Have evaluable disease per modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for immune based therapeutics (iRECIST).
* Have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1.
* Adequate bone marrow function, with absolute neutrophil count >1,500/µL, platelet count >75,000/µL, and hemoglobin >9g/dL (or 5.6 mmol/L).
* Adequate liver function with bilirubin <1.5 x the upper limit of normal (ULN) range, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x the ULN.
* Adequate renal function, as defined by having creatinine clearance ≥30 mL/min calculated by either Cockcroft-Gault or Modification of Diet in Renal Disease equations.
* Adequate cardiac function, no clinically significant abnormalities assessed by electrocardiogram (ECG), and absence of significant cardiac disease.
* Negative serum pregnancy test within 24 hours prior to start of study drug in female patients of childbearing potential. Not applicable to patients unable to become pregnant, including those with bilateral oophorectomy and/or hysterectomy or postmenopausal.
* Patients of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) during heterosexual intercourse, starting at screening and continuing throughout study, for a total of 31 weeks post-treatment completion.

Exclusion Criteria:

* Have ongoing toxicities >Grade 1 according to NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v5.0 (excluding alopecia and neuropathy).
* Have any contraindications to receiving cetuximab therapy, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 (anti-cytotoxic T-lymphocyte antigen) antibody, or other antibody or drug targeting T-cell co-stimulation or immune checkpoint pathways.
* Have known hypersensitivity to study drugs.
* Have undergone surgery and not recovered adequately from toxicities and/or complications from the intervention prior to starting study therapy; or have unresolved toxicity from prior radiation, chemotherapy, or other targeted treatment, including investigational treatment.
* Have clinically significant cardiac arrhythmia, unless well-controlled.
* Have clinically active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain or meningeal metastasis may participate and be eligible for treatment provided they are stable and asymptomatic, and have no evidence of new or enlarging brain metastases evaluated within 4 weeks prior to the first dose of study drug.
* Patients with history of human immunodeficiency virus (HIV) and:

  1. CD4+ T-cell count is ≤350 cells µL;
  2. History of AIDS-defining opportunistic infection within the past 12 months;
  3. Antiretroviral therapy <4 weeks and HIV viral load >400 copies/mL.
* Have participated in another investigational drug or device study within 4 weeks of the first dose of study drug.
* Female patient who is pregnant or breast feeding.
* Have signs or symptoms of organ failure, major chronic illnesses other than cancer, or any concomitant medical or social condition that, in the opinion of the investigator, make it undesirable for the patient to participate in the study, or that could jeopardize compliance with the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of dose-limiting toxicities (DLTs) | Up to Day 28
  Incidence of DLTs with single agent SYN125
Part B: Incidence of dose-limiting toxicities (DLTs) | Up to Day 28
  Incidence of DLTs with SYN125 and fixed-dose SYN004 administered in combination

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to Day 50
  Incidence of Adverse Events (AEs)
Incidence of Clinical Laboratory Abnormalities | Up to Day 50
  Defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)
Serum concentration time profiles (Area under the serum concentration-time curve from time zero to the last measurable concentration) | Up to Day 106
  Serum concentration time profiles (Area under the serum concentration-time curve from time zero to the last measurable concentration) of SYN125 and SYN004
Area under the serum concentration time-curve over the dosing interval | Up to Day 106
  Area under the serum concentration time-curve over the dosing interval of SYN125 and SYN004
Area under the serum concentration-time curve from time zero extrapolated to infinity (AUC0-inf) | Up to Day 106
  Area under the serum concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of SYN125 and SYN004
Maximum Observed Plasma Concentration (Cmax) | Up to Day 106
  Maximum Observed Plasma Concentration (Cmax) of SYN125 and SYN004
Time to maximum observed serum concentration (Tmax) | Up to Day 106
  Time to maximum observed serum concentration (Tmax) of SYN125 and SYN004
Terminal elimination half-life (t1/2) | Up to Day 106
  Terminal elimination half-life (t1/2) of SYN125 and SYN004
Clearance | Up to Day 106
  Clearance of SYN125 and SYN004
Volume of distribution at steady-state (Vss) | Up to Day 106
  Volume of distribution at steady-state (Vss) of SYN125 and SYN004

CONTACTS AND LOCATIONS:
Overall Officials: Ding Wang, MD, Principal Investigator — Henry Ford Hospital
Locations (4):
- United States (4):
  - University of Kansas Cancer Center, Clinical Research Center, 4350 Shawnee Mission Parkway, MS 6004, Fairway, Kansas
  - Henry Ford Health System, Henry Ford Hospital, Brownstown, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Oklahoma, Peggy and Charles Stephenson Cancer Center, 800 Northeast 10th Street, Oklahoma City, Oklahoma

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm